CLINICAL TRIAL: NCT00863863
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fed, Bioequivalence Study Of Griseofulvin 125 mg/5 mL Suspension Versus Grifulvin V® 125 mg/5 mL Suspension In Normal, Healthy, Non-Smoking Male And Female Subjects
Brief Title: A Relative Bioavailability Study of Griseofulvin 125 mg/5 mL Suspension Under Non-fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Christine Winslow, Director of Clinical Development, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3155
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Griseofulvin; Healthy subjects
MeSH Terms: interventions — Griseofulvin; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Griseofulvin 125 mg/5 mL Suspension, single dose
  Interventions: Drug: Griseofulvin 125 mg/5 mL Suspension, single dose
- B (Active Comparator): Grifulvin V® 125 mg/5 mL Suspension, single dose
  Interventions: Drug: Grifulvin V® 125 mg/5 mL Suspension, single dose

INTERVENTIONS:
Drug: Griseofulvin 125 mg/5 mL Suspension, single dose — A: Experimental Subjects received Alpharma formulated products under non-fasting conditions
  Other Names: Griseofulvin
  Arms: A
Drug: Grifulvin V® 125 mg/5 mL Suspension, single dose — B: Active comparator Subjects received Ortho Neutrogena formulated products under non-fasting conditions
  Other Names: Griseofulvin
  Arms: B

SUMMARY:
To compare the rate and extent of absorption of griseofulvin from a test formulation of Griseofulvin 125 mg/5 mL Suspension versus the reference Grifulvin V® 125 mg/5 mL Suspension under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: A randomized, two-way crossover, open-label, single-dose, fed design.

Official Title: A TWO-WAY CROSSOVER, OPEN-LABEL, SINGLE-DOSE, FED, BIOEQUIVALENCE STUDY OF GRISEOFULVIN 125 mg/5 mL SUSPENSION VERSUS GRIFULVIN V® 125 mg/5 mL SUSPENSION IN NORMAL, HEALTHY, NON-SMOKING MALE AND FEMALE SUBJECTS

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male or female with a minimum age of 18 years.
2. Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 29.9 kg/m2.
3. Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats/minute, temperature between 35.8°C and 37SC).
4. Negative for drugs of abuse and nicotine.
5. Negative for hepatitis B-surface antigen, hepatitis C and HIV.
6. Female subjects: negative for pregnancy (as evaluated by serum β-CG test).
7. No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides that they are not clinically significant.
8. Female subjects who are surgically sterile for at least 6 months or post-menopausal for at least 1 year, or who will avoid pregnancy for at least 10 days before the study, during the study and up until 1 month after the end of the study.
9. Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed ICF.

Exclusion Criteria:

1. Known history of hypersensitivity to griseofulvin (e.g. Grifulvin V®, gris-PEG®, Fulvicin®) penicillin, or drugs derived from the same species of Penicillium.
2. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless deemed not clinically significant by the Principal Investigator or Sub-investigator.
3. Presence of any significant physical or organ abnormality.
4. Any history or evidence of psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator or Sub-investigator.
5. History of presence of any skin conditions (e.g. dermatitis, eczema, psoriasis).
6. Presence of any skin rashes.
7. Any subject who has been previously diagnosed with porphyria.
8. Any clinically significant illness during the 4 weeks before this study.
9. Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
10. Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
11. Significant or recent history of asthma (after 12 years of age).
12. Any subject with a history of drug abuse.
13. Any subject with a recent (less than 1 year) history of alcohol abuse.
14. Use of any prescription medication within 14 days preceding this study.
15. Use of over-the-counter (OTC) medication within 7 days preceding this study (except for spermicidal/barrier contraceptive products).
16. Female subjects: use of contraceptives (oral, emergency [Plan B®], transdermal, implant, Mirena® IUD, NuvaRing®) within 30 days before drug administration or a depot injection of progestogen drug (e.g. Depo-Provera®) within 1 year before drug administration.
17. Female subjects: evidence of pregnancy or lactation.
18. Any subject who has had blood drawn within 56 days preceding this study, during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
19. Participation in a clinical trial with an investigational drug within 30 days preceding this study.
20. Any subject who has donated blood within 56 days preceding this study.
21. Any subject who has participated as a plasma donor in a plasmapheresis program within 7 days preceding this study.
22. Any subject who has adhered to a significantly abnormal diet during the 4 weeks preceding the first dose of the study.
23. Intolerance to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y. Tam,, MD, Principal Investigator — Biovail Contract Research
Locations (1):
- Biovail Contract Research (A Division of Biovail Corporation), Toronto, Ontario, Canada